CLINICAL TRIAL: NCT04586647
Title: Investigation of Healthy Eating Habits and Attitudes Toward Food During a Weight Loss Intervention
Brief Title: Attitudes Toward Food During a Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noom Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00046455
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Weight Loss; Overweight and Obesity; Overweight or Obesity; Eating Behavior; Food Habits; Eating Disorder Symptom
MeSH Terms: conditions — Obesity; Weight Loss; Overweight; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noom Health Weight Program (Experimental)
  Interventions: Behavioral: Noom Healthy Weight; mobile behavior change program for weight loss.
- Wait List Control (No Intervention)

INTERVENTIONS:
Behavioral: Noom Healthy Weight; mobile behavior change program for weight loss. — The intervention consists of a curriculum, provided through daily articles that users are encouraged to read; logging features for weight, meals, and physical activity; in-app groups; and a virtual coach, who will communicate with participants via in-app messaging. During the first week of the study, participants will be introduced to the program, the Noom app, and their coach.
  Coaches will use a secure dashboard to monitor patient progress, which is used to increase engagement and motivation. Participants are encouraged to log their weight and physical activity on a weekly basis, and meals daily.
  Arms: Noom Health Weight Program

SUMMARY:
The purpose of this study is to evaluate whether the Noom Healthy Weight Program, a digital behavior change weight loss intervention, creates a positive relationship with food, compared to a waitlist control group.

DETAILED DESCRIPTION:
This is a prospective randomized, controlled pilot study evaluating relationships towards food in overweight and obese Noom Healthy Weight participants.

Participants will be randomly assigned to one of two conditions (intervention, waitlist control). In the intervention condition, participants will have immediate access to the full Noom program after consenting to Noom's Research Policy, which states the collection of in app user data for research purposes. In the waitlist control condition, participants will be informed that they are on a waiting list and will be provided access to the full Noom program after 4 months after consenting to Noom's Research Policy.

Noom will have access to participants' username and email address. Before the start of the program, participants in both conditions will be emailed a survey containing the validated questionnaires mentioned below. The survey will also ask for demographic information such as race, ethnicity, and socioeconomic status. Survey responses will be linked to weight data by email address, but all data will be de-identified prior to analysis. The same survey, without demographic questions, will be sent to participants again at program end (4 months).

The intervention consists of a curriculum, provided through daily articles that users are encouraged to read; logging features for weight, meals, and physical activity; in-app groups; and a virtual coach, who will communicate with participants via in-app messaging. During the first week of the study, participants will be introduced to the program, the Noom app, and their coach.

Coaches will use a secure dashboard to monitor patient progress, which is used to increase engagement and motivation. Participants are encouraged to log their weight and physical activity on a weekly basis, and meals daily.

The primary outcome of this study is to assess self-reported eating behaviors via the Three Factor Eating Questionnaire following a 4 month weight loss intervention (Noom Healthy Weight program).

Secondary outcomes assessing disordered eating habits and mindfulness will be measured via the Disordered Eating Attitude Questionnaire and the Mindful Eating Scale. Mean weight loss differences between groups will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide informed consent
* 18 years and older
* Self-report of good health
* Not diagnosed with an eating disorder
* Overweight or obesity (BMI ≥ 25)
* Able to meet our criteria of adherence to the program (at least 1 engagement per week on
* one of the following: logged exercise, logged meals, steps, weigh-ins, coach messages, read articles, and days with at least one weigh-in.) For females
* Not 6 months postpartum
* Not planning to become pregnant in the next 5 months.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent
* Currently pregnant or 6 months postpartum
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the quality of the data
* E.g., eating disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Self-reported eating behaviors via the Three Factor Eating Questionnaire | 4 months
  The primary outcome of this study is to assess self-reported eating behaviors via the Three Factor Eating Questionnaire following a weight loss intervention This assessment is designed to measure 3 dimensions of human eating behavior: cognitive restraint of eating (Factor I - 20 items), disinhibition (Factor II - 16 items), and hunger (Factor III - 15 items). The minimum score for factors I-II-III is therefore 0-0-0, and maximum possible score is 20-16-15. Part I includes items 1-36 and are rated either 1-True or 0-False. Part II includes items 37-51 and is rated on a 4-point scale with the exception of item 50, which is rated on a 6-point scale.
  Higher scores reflective of higher restraint,

SECONDARY OUTCOMES:
Self reported disordered eating habits via the Disordered Eating Attitude Questionnaire | 4 months
  A 25-item questionnaire that assesses the individual's eating attitudes.
Self reported mindful eating habits via the Mindful Eating Scale | 4 months
  self-report scale to measure mindfulness with respect to eating behaviors

CONTACTS AND LOCATIONS:
Locations (1):
- Noom, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No